CLINICAL TRIAL: NCT00927030
Title: Melatonin for Sleep in Children With Autism: Safety Tolerability and Dose
Brief Title: Melatonin for Sleep in Children With Autism
Acronym: NICHD
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vanderbilt University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Beth Ann Malow, Professor, Departments of Neurology and Pediatrics, Vanderbilt University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 071269
Record Dates: First submitted 2009-06-22; First posted 2009-06-24 (Estimated); Last update posted 2012-07-02 (Estimated); Status verified 2012-06

CONDITIONS: Autistic Disorder; Insomnia
Keywords: Autism; children; sleep; insomnia
MeSH Terms: conditions — Autistic Disorder; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pharmacokinetic (Experimental): We hope to target 12 of the 30 children to be enrolled for this study to participate in a pharmacokinetic arm of the study. These 12 children would be receiving overnight sleep studies prior to receiving the first dose of melatonin and again at about every 3 week intervals each time the dose increases until the child is falling asleep within 30 minutes of bedtime on 5/7 nights per week. During the sleep studies an intravenous catheter will be placed in the child's arm to sample small amounts of blood throughout the day (about 3 teaspoons of blood)to allow us to look at how melatonin is produced in children with autism who have sleep problems.
  Interventions: Drug: supplemental liquid melatonin
- flavored inert liquid (Placebo Comparator): Of the 30 targeted participants, 18 will be randomized at the first three week dosing period {1mg of melatonin}. The randomization will be single blind to the parent in a 5:1 ratio (15 children will receive melatonin, and 3 children will receive a flavored placebo at the first 3-week period only). After the initial 3-week dose cycle of 1 mg, all children randomized to placebo will begin 3 mg of melatonin and will continue in dose increase (6mg, 9 mg)until they meet the criteria of falling asleep within 30 minutes of bedtime 5/7 nights per week. No child will take more than 9 mg.
  Interventions: Drug: flavored liquid or liquid supplemental melatonin

INTERVENTIONS:
Drug: supplemental liquid melatonin — Liquid melatonin will be given to the parent. There are 4 dose levels (1mg, 3mg, 6 mg, and 9mg)of melatonin that will be used at 3 week intervals. The child will start with 1mg and the dose will be increased at 3 week intervals until the child is falling asleep within 30 minutes of bedtime on 5/7 nights per week. Once this goal is reached the child will stay on that dose through the remainder of the study.
  Other Names: Natrol brand liquid melatonin
  Arms: Pharmacokinetic
Drug: flavored liquid or liquid supplemental melatonin — Single blind for parents at initial 3-weeks dose period of 1 mg melatonin for 18 children where 3/18 children will receive placebo and 15/18 children will receive melatonin study drug. Each bottle will be labeled as: Flavored liquid placebo/or liquid melatonin. After this initial 3-week period all children will receive known melatonin in bottles that state this.
  Other Names: Inert flavored liquid manufactored by PharmaCare in Mt. Juliet TN. A certificate of analysis is on file for this compounded liquid.
  Arms: flavored inert liquid

SUMMARY:
The purpose of this study is to determine if liquid supplemental melatonin is an effective treatment for children with autism who have sleep problems related to insomnia (difficulty falling asleep).

DETAILED DESCRIPTION:
Sleep difficulties in children with autism spectrum disorders (ASD) are common reasons why parents seek medical intervention for their children. Identifying a safe and effective pharmacologic agent that promotes sleep in ASD would favorably impact the lives of these children and their families. In this study we plan to determine the dose-response, tolerability and any adverse effects of supplemental melatonin in 30 children with ASD.The melatonin dose levels are 1mg, 3mg, 6mg, and 9mg. After a 3 week baseline period, the child will begin melatonin at 1mg and will dose escalate every three weeks until he/she is falling asleep within 30 minutes of bedtime at least 5/7 nights per week. No child will take more than 9 mg of supplemental melatonin.

ELIGIBILITY:
Inclusion Criteria:

* Children with autism ages 4-10 years.
* Diagnosis of autism based on Autism Diagnostic Observation Schedule (ADOS).
* Time to fall asleep of 30 minutes or longer by parent report at least 3 nights/week in the last 3 months.
* Children may take seasonal allergy medications.
* Children may take the following medications for the same dose at least 3 months: Citalopram (Celexa), Escitalopram (Lexapro), Amphetamine-dextroamphetamine (Adderall), Atomoxetine (Strattera), Methylphenidate(Ritalin), Dextroamphetamine(Dexedrine), Risperidone (Risperdal.

Exclusion Criteria:

* Children taking medications other than those in the inclusion criteria.
* Children with primary sleep disorder other than insomnia (such as sleep-disordered breathing).
* Children with non-febrile unprovoked epileptic seizure within the last two years.
* Children with liver disease or high fat diets, as melatonin metabolism may be affected in these children.
* Children who are visually impaired (partially or completely blind) as light suppresses melatonin synthesis and these children may have altered diurnal melatonin rhythms.
* Children with known genetic syndromes co-morbid with autism including fragile X, Down syndrome, neurofibromatosis, or tuberous sclerosis.
* Children who have outside normal limits on blood work for complete blood count, liver and renal function and hormone levels of ACTH, cortisol, LH, FSH, prolactin, testosterone and estradiol.
* Tanner staging beyond level 1 at any time point in the study.
* Children whose assessment score does not place them on the autism spectrum.

Ages: 4 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 17 (Actual)
Dates: Start 2008-01; Primary Completion 2010-04 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Determine dose-response, tolerability, and adverse effects of melatonin in 30 children with autism. | Two Years from study start

SECONDARY OUTCOMES:
A sub-set of 12 children will be studied to characterize the pharmacokinetic profile of orally administered melatonin. | 2 years from start of study
A group of behavioral and parental stress measures will be piloted for the participants in this study. | 2 years from start of study

CONTACTS AND LOCATIONS:
Overall Officials: Beth A Malow, MD, MS, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt Medical Center, Nashville, Tennessee, United States